CLINICAL TRIAL: NCT00243412
Title: A Double-Blind, Randomized, Multicenter, Phase II Study of the Safety and Efficacy of Two Rituximab Regimens in Subjects With Moderate to Severe Active Rheumatoid Arthritis Receiving Stable Doses of Methotrexate
Brief Title: A Study of the Safety and Efficacy of Rituximab in Patients With Moderate to Severe Rheumatoid Arthritis Receiving Methotrexate
Acronym: RUMBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U3377g
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituxan; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; Methotrexate; Methylprednisolone; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A: 500 mg Rituximab (Experimental): Rituximab: 1000 mg intravenous (IV) on Days 1 and 15 of the first cycle; 500 mg IV on Days 1 and 15 of each subsequent 6-month cycle (Months 6, 12, and 18).
  Corticosteroids: 100 mg IV methylprednisolone prior to each rituximab infusion.
  Methotrexate: 15-25 mg/wk oral or parenteral (10-14 mg/wk if intolerant).
  Folate: Minimum of 1 mg/day (or folinic acid 5 mg/wk).
  Interventions: Drug: folate; Drug: methotrexate; Drug: methylprednisolone; Drug: Rituximab
- Arm B: 1000 mg Rituximab (Experimental): Rituximab: 1000 mg IV on Days 1 and 15 of each 12-month cycle (Rituximab cycles were administered at baseline and Month 12.) For the Month 6 and 18 cycles, rituximab or placebo was administered.
  Corticosteroids: 100 mg IV methylprednisolone prior to each rituximab infusion For the Months 6 and 18 cycles, IV saline was administered prior to each rituximab or placebo infusion.
  Methotrexate: 15-25 mg/wk oral or parenteral (10-14 mg/wk if intolerant).
  Folate: Minimum of 1 mg/day (or folinic acid 5 mg/wk).
  Interventions: Drug: folate; Drug: methotrexate; Drug: methylprednisolone; Drug: Placebo; Drug: Rituximab

INTERVENTIONS:
Drug: folate — Minimum of 1 mg/day oral (or folinic acid 5 mg/week)
Drug: methotrexate — 15-25 mg/week oral or parenteral (10-14 mg/week if intolerant)
Drug: methylprednisolone — 100 mg intravenous (IV) prior to each rituximab infusion (For Arm B, for the Months 6 and 18 cycles, IV saline was administered prior to each placebo infusion)
Drug: Placebo — To maintain the blind, patients in Arm B (Rituximab 1000 mg) received placebo infusions at Months 6 and 18.
  Arms: Arm B: 1000 mg Rituximab
Drug: Rituximab — 500 mg or 1000 mg IV*2.

SUMMARY:
This was a Phase II, randomized, double-blind, multicenter study designed to evaluate the safety and efficacy of rituximab, administered at two different regimens for 2 years, in patients with moderate to severe active rheumatoid arthritis (RA) receiving stable doses of methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for at least 6 months.
* Inadequate response to MTX
* Use of folate
* If female and of childbearing potential, have a negative serum pregnancy test within 8 weeks prior to first rituximab infusion

Exclusion Criteria:

* Diagnosis of juvenile idiopathic arthritis (also known as juvenile rheumatoid arthritis) and/or RA before age 16
* Any surgical procedure, including bone/joint surgery or planned surgery within 8 weeks prior to screening or within 16 weeks of Week 1 (Day 1) visit
* Inflammatory arthritis other than RA (e.g., inflammatory bowel disease, systemic lupus erythematosus (SLE), or psoriatic arthritis)
* Functional Class IV as defined by the American College of Rheumatology (ACR) classification of functional status in RA
* Use of disease-modifying anti-rheumatic drugs (DMARDs) other than MTX within 4 weeks prior to randomization (8 weeks prior for infliximab, adalimumab, or leflunomide)
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Previous treatment with Tysabri<TM> (natalizumab)
* Previous treatment with rituximab
* Previous treatment with any cell-depleting therapies, including investigational agents
* Treatment with IV &-globulin or Prosorba(R) Column within the previous 6 months
* Use of intra-articular or parenteral corticosteroids within 4 weeks prior to screening visit
* Receipt of a vaccine within 4 weeks prior to Day 1 infusion
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Primary or secondary immunodeficiency (history of or active)
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, renal, hepatic, endocrine, gastrointestinal, or pulmonary disease, including any pulmonary or other condition that would preclude subject participation over the ensuing 2 years
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds)
* History of recurrent significant infection or any significant episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* History of significant cytopenias or other bone marrow disorders
* History of cancer, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinoma of the skin that have been excised and cured)
* Pregnant or nursing (breast feeding) women
* Lack of peripheral venous access
* Chronic daily use of narcotic analgesics
* History of alcohol, drug, or chemical abuse within 6 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Reiss, Pharm.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 40 subjects with moderately to severely active rheumatoid arthritis were to be enrolled at six to eight study centers in the United States and were randomly assigned in a 1:1 ratio to Arm A or B. Starting 15 August 2005 to 4 February 2009 (first subject enrolled to database lock).
Pre-assignment Details: All subjects were to receive rituximab 1000 mg * 2 on Days 1 and 15. Subsequently, subjects in Arm A received rituximab 500 mg * 2 every 6 months (Months 6, 12, and 18) and those in Arm B received rituximab 1000 mg * 2 at 12 months. To maintain the blind, subjects in Arm B received placebo infusions at Months 6 and 18.
Groups:
- Arm B: 1000 mg Rituximab: Rituximab: 1000 mg IV on Days 1 and 15 of each 12-month cycle (Rituximab cycles were administered at baseline and Month 12). For the Month 6 and 18 cycles, rituximab or placebo was administered. Corticosteroids: 100 mg IV methylprednisolone prior to each rituximab infusion, For the Months 6 and 18 cycles, IV saline was administered prior to each rituximab or placebo infusion. Methotrexate: 15-25 mg/wk oral or parenteral (10-14 mg/wk if intolerant). Folate: Minimum of 1 mg/day (or folinic acid 5 mg/wk).
Period: Overall Study
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Started | 21 (Intent to treat) | 21 (Intent to treat)
Safety Evaluable | 21 | 20
Completed | 11 (Completed Week 104) | 10 (Completed Week 104)
Not Completed | 10 | 11
Not completed — Death | 0 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: 500 mg Rituximab: Rituximab: 1000 mg IV on Days 1 and 15 of the first cycle; 500 mg IV on Days 1 and 15 of each subsequent 6-month cycle (Months 6, 12, and 18). Corticosteroids: 100 mg IV methylprednisolone prior to each rituximab infusion. Methotrexate: 15-25 mg/wk oral or parenteral (10-14 mg/wk if intolerant). Folate: Minimum of 1 mg/day (or folinic acid 5 mg/wk).
- Arm B: 1000 mg Rituximab: Rituximab: 1000 mg IV on Days 1 and 15 of each 12-month cycle (Rituximab cycles were administered at baseline and Month 12). For the Month 6 and 18 cycles, rituximab or placebo was administered. Corticosteroids: 100 mg IV methylprednisolone prior to each rituximab infusion. For the Months 6 and 18 cycles, IV saline was administered prior to each rituximab or placebo infusion. Methotrexate: 15-25 mg/wk oral or parenteral (10-14 mg/wk if intolerant). Folate: Minimum of 1 mg/day (or folinic acid 5 mg/wk).
- Total: Total of all reporting groups
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 46.9 (9.6) | 47.4 (11.1) | 47.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Either an Infection or a Grade III or IV Adverse Event (National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI CTCAE], Version 3.0)
Description: A Grade III Adverse Event (AE) is severe; defined as considerable interference with the subject's daily activities, medical intervention/therapy required and hospitalization possible.
  A Grade IV AE is life-threatening; defined as extreme limitation in activity, significant medical intervention/therapy required, hospitalization probable.
  Because of the small sample size and the small number of subjects who completed Week 104, the analysis were limited to descriptive statistics only.
Time Frame: 24 months
Population: Safety-Evaluable Population
Measure: Number; unit: Participants
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 21 | 20
Participants
  Infections | 14 | 11
  Adverse Events (Grade 3 or 4) | 5 | 4

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28-4 C-reactive Protein (DAS28-4(CRP))
Description: The DAS28-4(CRP) score is a measure of the subject's disease activity. DAS28-4(CRP) is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity and CRP. DAS28 provides a number on a scale (0 to 10) indicating current disease activity. A score above 5.1 means high disease activity and a score below 3.2 indicates low disease activity. Change from baseline at 24 months was analyzed for DAS28-4 (CRP).
Time Frame: Baseline, 24 months
Population: Participants from the Intent-to-Treat (ITT) population for whom data was available at baseline and month 24.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
Scores on a scale
  Baseline | 6.53 (0.70) | 6.33 (0.85)
  Month 24 | 4.03 (1.75) | 3.77 (1.42)
  Change from baseline | -2.49 (1.85) | -2.56 (1.23)

3. Secondary Outcome: Number of Participants With American College of Rheumatology Responses (ACR20, ACR50, and ACR70)
Description: ACR20 response was defined as satisfying the following 3 criteria improvement from baseline: ≥ 20% in tender joint count; ≥ 20% in swollen joint count; ≥ 20% improvement from baseline in 3 of the following 5 criteria:
  Subject's Global Assessment of Pain Subject's Global Assessment of Disease Activity Physician's Global Assessment Subject's Self-Assessment Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP) Note: The definitions of ACR50 and ACR70 are the same as ACR20, except that the 20% value in the above definition is replaced by 50% and 70% values, respectively.
Time Frame: Baseline, 24 months
Population: Intent-to-Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 21 | 21
Participants
  ACR20 Responders | 7 | 6
  ACR50 Responders | 4 | 5
  ACR70 Responders | 4 | 3

4. Secondary Outcome: Number of Participants With American College of Rheumatology (ACR) Major Clinical Response and/or Remission
Description: Major clinical response is an ACR70 response defined as improvement from baseline: ≥70% in tender joint count; ≥70% in swollen joint count; ≥70% in 3 of the following: Patient Pain Assessment, Patient Global Assessment, Physician Global Assessment, Patient Self-Assessed Disability, ESR or CRP for ≥169 consecutive days.
  Remission: ≥5 requirements fulfilled for ≥2 consecutive months: Duration of morning stiffness <15 minutes, No fatigue, No joint pain, No joint tenderness or pain on motion, No soft tissue swelling in joints or tendon sheaths, ESR <30 mm/hour for women and <20 mm/hour for men.
Time Frame: 24 months
Population: Intent-to-Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 21 | 20
Participants | 1 | 0

5. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response and Remission Using Disease Activity Score 28-4 (DAS28-4)C-reactive Protein (CRP)
Description: EULAR remission = DAS28-4(CRP) < 2.6 (Fransen et al. 2004.
  EULAR response categories (van Gestel et al. 1999):
  Good response = final DAS28-4(CRP) < 3.2 and decreased > 1.2 points from baseline Moderate response = final DAS28-4(CRP) ≥ 3.2 but ≤ 5.1 and decreased > 0.6 points from baseline or final DAS28-4(CRP) > 5.1 and decreased > 1.2 from baseline.
Time Frame: Baseline, 24 months
Population: Participants from the Intent-to-Treat (ITT) population for whom data was available at baseline and month 24.
Measure: Number; unit: Participants
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
Participants
  No Response | 0 | 0
  Moderate Response | 2 | 6
  Good Response | 5 | 4
  Eular Remission | 3 | 3

6. Secondary Outcome: Change From Baseline in Short Form 36 (SF 36) Summary and Subscale Scores
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning (PF), Role Physical (RP), Bodily Pain(BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE),Mental Health (MH). Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score.
Time Frame: Baseline, 24 Months
Population: Participants from the Intent-to-Treat (ITT) for whom data was available at baseline and month 24.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
Units on a Scale
  Summary Score: Mental Component Score | 7.69 (16.10) | 2.28 (10.42)
  Summary Score: Physical Component Score | 9.88 (12.31) | 4.93 (9.83)
  Subscale: Bodily Pain | 26.64 (26.64) | 8.00 (22.55)
  Subscale: General Health | 13.86 (18.78) | 18.40 (23.55)
  Subscale: Mental Health | 20.00 (18.17) | 2.50 (26.48)
  Subscale: Physical Function | 21.62 (35.45) | 15.72 (17.54)
  Subscale: Role Emotional | 16.67 (45.95) | 8.33 (24.85)
  Subscale: Role Physical | 34.09 (31.17) | -1.25 (23.90)
  Subscale: Social Functioning | 21.59 (35.83) | 7.50 (25.14)
  Subscale: Vitality | 10.61 (26.03) | 8.13 (12.86)

7. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The Stanford HAQ-DI is a patient-reported questionnaire specific for RA. It consists of 20 questions referring to eight component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. The questionnaire was provided in a certified translation of the local languages at the participating sites and was scored based on the instructions from the Stanford University Medical Center.The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction.
Time Frame: Baseline, 24 Months
Population: Participants from the Intent-to-Treat (ITT) population for whom data was available at baseline and month 24.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
Scores on a scale | -0.60 (0.87) | -0.45 (0.72)

8. Secondary Outcome: Change From Baseline in Functional Assessment for Chronic Illness Therapy-Fatigue (FACIT-F)
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the patient's health status.
Time Frame: Baseline, 24 Months
Population: Participants from the Intent-to-Treat (ITT) population for whom data was available at baseline and month 24.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
Scores on a scale | 9.64 (15.54) | 8.80 (12.15)

9. Secondary Outcome: DAS28-4 Erythrocyte Sedimentation Rate(ESR)
Description: The DAS28-4(ESR) score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR. DAS28-4(ESR) scores range from 0 - 10, where a score of less than or equal to 3.2 implies well controlled disease and greater than or equal to 5.1 implies active disease In this trial, CRP rather than ESR was used, unless the CRP value was missing at both Day 1 and screening, in which case ESR value was used.
Time Frame: 24 Months
Population: Participants from the Intent-to-Treat (ITT) for whom data was available at baseline and month 24.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
Scores on a scale | 4.25 (1.98) | 4.32 (1.39)

10. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF)
Description: Serum levels of rheumatoid factor at baseline, month 24 and change from baseline to month 24.
Time Frame: Baseline, 24 Months
Population: Participants from the Safety-Evaluable population for whom data was available at baseline and month 24.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 11 | 10
IU/mL
  Baseline | 542.8 (1011.6) | 243.7 (280.2)
  Month 24 | 43.0 (70.8) | 41.4 (34.3)
  Change from Baseline to Month 24 | -499.8 (946.9) | -202.3 (279.1)

11. Secondary Outcome: Change From Baseline in Cyclic Citrullinated Peptide (CCP) Antibodies/Cytokines
Description: Because of the different laboratory methods that were used to measure anti-CCP antibody levels, no summary statistics were calculated.
Time Frame: Baseline, 24 Months
Measure: Number; unit: units
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration includes safety-evaluable subjects during the 2-year treatment period; in addition Serious adverse events that occurred during safety follow-up.
Description: A total of 42 subjects were randomized into the trial, 21 in Group A (500 mg rituximab retreatment regimen) and 21 in Group B (1000 mg rituximab retreatment regimen). Twenty subjects in Group B were treated with study drug and included in the safety-evaluable population.
Arm/Group | Arm A: 500 mg Rituximab | Arm B: 1000 mg Rituximab
Serious Adverse Events (participants affected / at risk) | 3/21 | 2/20
Other Adverse Events (participants affected / at risk) | 21/21 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 500 mg Rituximab (N=21) | Arm B: 1000 mg Rituximab (N=20)
DEATH (Cardiac disorders) | 0 | 1 — CARDIAC ARREST
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 500 mg Rituximab (N=21) | Arm B: 1000 mg Rituximab (N=20)
Nausea (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 7
Sinusitis (Infections and infestations) | 6 | 1
Urinary tract infection (Infections and infestations) | 2 | 3
Fungal infection (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 3 | 0
Liver function test abnormal (Investigations) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Insomnia (Nervous system disorders) | 4 | 3
Anxiety (Nervous system disorders) | 1 | 2
Depression (Nervous system disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis, allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 2 | 2
Hot flush (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Because of the limited sample size, interpretation of these results should be made with caution and therefore definitive conclusions cannot be made regarding differences between the two retreatment regimens studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.